CLINICAL TRIAL: NCT06897566
Title: Evaluation of Adherence to Cholesterol Therapies and Identification of Barriers to Optimal LDL-C Targets in Patients With Atherosclerotic Cardiovascular Disease
Brief Title: Barriers to Optimal LDL-C Targets in Patients With Atherosclerotic Cardiovascular Disease
Acronym: BOLT
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmad Samir, Professor, Cairo University
Other Study IDs: MS1462021
Record Dates: First submitted 2025-03-19; First posted 2025-03-27 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Statin Adverse Reaction; LDL Level
Keywords: coronary artery disease; LDL-C; statins; statin intolerance; statin associated muscle symptoms
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fasting lipid profile — Recruited patients will be requested to provide data from their most recent fasting lipid profile

SUMMARY:
In the present cross-sectional observational study, the investigators aimed to:

* Evaluate the prevalence of achievement of LDL-C targets among a sample of Egyptian ASCVD patients.
* Attempt to unveil the potential barriers to achieve LDL-C goals in order to determine the appropriate corrective actions.

DETAILED DESCRIPTION:
There is a huge gap between guideline recommendations and real-world data concerning LDL-C targets for coronary artery disease CAD patients. This large gap highlights the need to improve the utilization of high-intensity statins and other non-statin therapies. This dictates evaluating the reasons for underutilization of statin and non-statin therapies, as well as understanding the barriers to achieving optimal LDL-C targets. Although there are few attempts to document and analyze this gap, all of them come from the Western world while data from the Middle East are sparse.

This cross-sectional observational study to evaluate the prevalence of achievement of LDL-C targets among a sample of Egyptian CAD patients. Also potential barriers to LDL-C goals will be sought in order to determine the appropriate corrective actions.

- Population of study: Patients with ASCVD and eligible for high-intensity statin therapy for a period of 6-months or more.

- Study location: Cairo University hospitals.

* Inclusion criteria:
* Patients presenting to cardiology department/ outpatient clinic.
* Established ASCVD and eligible for high intensity statins for at least six-months.
* Age between18-to-80y.
* Exclusion criteria:
* Refusal to participate in the survey.
* Patients with medical limitation or contraindications to statins therapy.
* Patients with documented diagnosis of homozygous familial hypercholesterolemia.
* Methodology in details:

Patients meeting the eligibility criteria will be offered to participate in the online survey tool through their smart phones. The link and the QR-code for the tool will be offered to the patient, and assistance will be offered to resolve any ambiguity of the questions if needed.

The patient would respond to the 38-item questionnaire comprising the study tool that can be accessed by their phones.

https://forms.office.com/r/xni4uNWKGg and a QR-code (can not be pasted to this text box) was available for swift and easy access.

Data were automatically pooled into an electronic online database for analysis upon study completion.

- Confidentiality of data: Clinical data will be tabulated by number codes that will be anonymized. Only treating physicians will have access to participants identities, while the anonymized tabulated data will be available for the statisticians.

* Study outcomes:
* Primary outcome parameters Prevalence of achievement of recommended LDL-C targets among patients with established ASCVD.
* Secondary outcome parameters Identify potential barriers to achieve LDL-C targets.
* Sample size This survey is planned to be completed when 1000 ASCVD patients finish their participation to the online survey tool.
* Statistical analysis Statistical package for social science (SPSS) software, version 22 for Microsoft Windows (SPSS Inc., Chicago, IL, USA) will be used for data analysis. Categorical data will be presented as frequency and percentages (n (%)) and correlations among them will be analyzed by chi square test. Continuous data will be checked for normality using Shapiro-Wilk test and will be presented as mean (standard deviation) or median (interquartile range) as appropriate. Continuous data will be analyzed using one-way analysis of variance (ANOVA). Repeated measures will be analyzed using analysis of variance (ANOVA) for repeated measures with post-hoc pairwise comparisons using the Tukey and Bonferroni tests. A probability p value less than 0.05 will be considered statistically significant.
* Source of funding:
* None

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to cardiology department/ outpatient clinic.
* Established ASCVD and eligible for high intensity statins for at least six-months.
* Age between18-to-80y.

Exclusion Criteria:

* Refusal to participate in the survey.
* Recent diagnosis of ASCVD with indication to high intensity statins for a period < six-months.
* Patients with medical limitation or contraindications to statins therapy.
* Patients with documented diagnosis of homozygous familial hypercholesterolemia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with established ASCVD with indication for high-intensity statin for a period 6 months This includes patients with coronary artery disease, peripheral arterial disease, cerebrovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2024-09-21 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of achievement of recommended LDL-C targets among patients with established ASCVD | Being a cross sectional study selectively recruiting patients with established indication for >6months, the study will accept a fasting lipid profile that was performed within 1 month from surveying the recruited patient.
  Recruited patients will be stratified according to the LDL-C levels into those <55, <70, <100, <130, and above.
  Patients in different LDL-C strata will be surveyed. Predictors for failure of achievement of LDL-C goals will be sought.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Medicine Cairo University, Cairo
  - Faculty of Medicine, Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided